CLINICAL TRIAL: NCT06259825
Title: Omega-3-Index Response to Eating Poultry Foods Naturally Enriched With Omega-3 Polyunsaturated Fatty Acids: A Randomized Controlled Trial in Healthy Saudi Adults
Brief Title: Omega-3-Index Response to Eating Poultry Foods Naturally Enriched With Omega-3 Polyunsaturated Fatty Acids
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King Abdulaziz University (Other)
Collaborators: Royal College of Surgeons, Ireland (Other); University College Dublin (Other)
Responsible Party: Principal Investigator, Salwa Ali Albar, Associate Professor, King Abdulaziz University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: KAU-664-23
Record Dates: First submitted 2024-02-07; First posted 2024-02-14 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Healthy Nutrition; Healthy Adults
Keywords: Omega-3 Polyunsaturated Fatty Acids; Omega-3 PUFAs; Poultry Foods; Chicken-meat; Eggs; Randomized Nutritional Trial
MeSH Terms: interventions — Docosahexaenoic Acids; Eggs

STUDY DESIGN:
Intervention Model Description: This will be a randomised double-blind interventional study.
  Participants will be randomized to either of two arms;
  * Control / Placebo Intervention: Consumption of at least 4 portions of standard chicken-meat and at least 4 standard eggs per week, for 4 months.
  * Experimental Intervention: Consumption of at least 4 portions of omega-3-PUFA enriched chicken-meat and at least 4 omega-3-PUFA enriched eggs per week, for 4 months.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The randomization schedule was computer generated. Separate sealed opaque envelopes were prepared for male, female and couple participants. Participants and all investigators involved in participant recruitment, data collection and entry, sample collection, processing and analysis, will be masked to the randomization groups until data entry is completed and the database is locked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Chicken-meat and Control Eggs (Placebo Comparator): Consumption of at least 4 portions of standard chicken-meat and at least 4 standard eggs per week, for 4 months.
  Interventions: Other: Control poultry foods (chicken-meat and eggs)
- Omega-3 Chicken-meat and Omega-3 Eggs (Experimental): Consumption of at least 4 portions of omega-3-PUFA enriched chicken-meat and at least 4 omega-3-PUFA enriched eggs per week, for 4 months.
  Interventions: Other: Omega-3 polyunsaturated fatty acid, naturally enriched, poultry foods (chicken-meat and eggs)

INTERVENTIONS:
Other: Omega-3 polyunsaturated fatty acid, naturally enriched, poultry foods (chicken-meat and eggs) — At least four portions of omega-3 PUFA enriched chicken-meat (whole chickens, breasts, thighs and drums) and at least four omega-3 PUFA enriched eggs will be consumed weekly for 4 months. The poultry meat and eggs will be enriched by feeding chickens a complete feed which includes algae, which is a rich source of omega-3 PUFAs (OmegaPro, Humanitiv, Meath, Ireland).
  Arms: Omega-3 Chicken-meat and Omega-3 Eggs
Other: Control poultry foods (chicken-meat and eggs) — At least four portions of standard chicken-meat (whole chickens, breasts, thighs and drums) and at least four standard eggs will be consumed weekly for 4 months.
  Arms: Control Chicken-meat and Control Eggs

SUMMARY:
Diets low in seafood omega-3 polyunsaturated fatty acids (PUFAs) are very prevalent. Such diets have recently been ranked as the sixth most important dietary risk factor-1.5 million deaths and 33 million disability-adjusted life-years worldwide are attributable to this deficiency. Wild oily fish stocks are insufficient to feed the world's population, and levels of eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA) in farmed fish have more than halved in the last 20 years.

The primary objective of this randomised, double-blinded, controlled nutritional trial will be to test if consumption of at least 4 servings of omega-3 PUFA-enriched chicken-meat and 4 enriched eggs per week, over a 4-month period, results in measurably higher blood levels of EPA and DHA in healthy Saudi adults.

This will be a randomised double-blind interventional study. Eighty adult male and female participants (age ≥ 18 years of age) will be asked to eat at least 4 portions of omega-3-PUFA enriched (or control) chicken-meat per week, and at least 4 omega-3-PUFA enriched (or control) eggs per week, for 4 months. Participants will be assessed at baseline and at monthly intervals for 4 months. Assessments at these visits will include; comprehensive lifestyle and medical history; food frequency questionnaire; 3 days food record; height, weight, waist and hip circumferences; blood sampling; participant well-being and adverse events. Measurement of plasma and red blood cell levels of EPA, DHA and Docosapentaenoic acid (DPA) will be performed at baseline and at study end using gas chromatography-mass spectroscopy.

The primary end point will be the change in red blood cell omega-3-index (sum of EPA and DHA expressed as percentage of total fatty acids in erythrocyte membranes) at 4 months. The nutritional trial will be analyzed on an intension to treat basis. Repeated measures ANOVA will be used to compare the two study groups. The study will be reported in accordance with the CONSORT (Consolidated Standards of Reporting Trials) 2010 statement.

DETAILED DESCRIPTION:
STUDY RATIONALE

In this randomized, double-blinded, controlled trial, the investigators aim to quantify the impact of regular consumption of omega-3 PUFA enriched chicken-meat and eggs over a four month period, in a healthy Saudi population.

STUDY AIMS AND OBJECTIVES.

The primary objective of this study will be to assess the red blood cell omega-3 index response of healthy Saudi adults to regular consumption of omega-3 PUFA-enriched chicken-meat and eggs. The red blood cell omega-3 index is calculated as the sum of EPA and DHA expressed as a percentage of total fatty acids in erythrocyte (red cell) membranes.

Secondary objectives include;

* The assessment of red cell and plasma EPA, DPA and DHA responses to regular consumption of omega-3 PUFA-enriched chicken-meat and eggs.
* The comparison of baseline red cell and plasma levels of EPA, DPA and DHA, amongst Saudi residents who regularly consume oily fish with those that do not regularly consume oily fish, and
* The assessment of whether the red cell and plasma omega-3 index responses to the omega-3-PUFA enriched foods differs between those that do, and those who do not, include oily fish in their weekly diet.

TRIAL DESIGN.

This will be a randomised double-blind interventional study. The trial will be performed in accordance with the Declaration of Helsinki.

STUDY PARTICIPANTS

80 healthy, community dwelling, participants will be recruited to the study.

RANDOMIZATION AND MASKING

Participants will be randomized to either of two arms;

* Control / Placebo Intervention: Consumption of at least 4 portions of standard chicken-meat and at least 4 standard eggs per week, for 4 months.
* Experimental Intervention: Consumption of at least 4 portions of omega-3-PUFA enriched chicken-meat and at least 4 omega-3-PUFA enriched eggs per week, for 4 months.

STUDY CONDUCT

Participants will attend the study center at the screening and baseline visits and at study end (month 4). They will be contacted by telephone at monthly intervals (Months 1, 2 and 3).

At the screening visit, a comprehensive lifestyle and medical history will be taken, a food frequency questionnaire will be completed to capture food intake over the previous year; a 3 days food record will be arranged to capture the current dietary intake of participants; and satisfaction of the inclusion and exclusion criteria will be evaluated.

At the baseline visit, if all inclusion and exclusion criteria are satisfied, participants will be randomized to either the control or the interventional arm of the study.

At both the baseline and month 4 visits, height, weight, waist and hip circumference will be measured, allowing calculation of both the body mass index and the waist-hip ratio. At these two clinic visits fasting blood samples will be taken to allow measurement of plasma and red cell levels of EPA, DPA and DHA, and also to allow storage of plasma aliquots for future research measurements. Participants will be asked to fast, not drink tea or coffee, not smoke and not engage in intense exercise from midnight (minimum 8 hours), prior to the baseline and end-of-study visits. Participants may drink water and take essential medications on these mornings.

At the month 1, 2 and 3 telephone calls, and at the month 4 visit, frequency of consumption of chicken-meat, eggs and fish, during previous week, will be assessed, as will concurrent medications and participant wellbeing.

Participants will be asked to avoid taking long-chain omega-3 PUFA supplements, for the duration of the study.

NUTRITIONAL INTERVENTION

The poultry meat and eggs will be enriched by feeding chickens a complete feed which includes algae, which is a rich source of omega-3 PUFAs (OmegaPro, Humanitiv, Meath, Ireland). Omega-3 PUFA enriched chicken (whole chickens, breasts, thighs and drums) and eggs, or the appropriate control chicken and control eggs, will be delivered to the homes of study participants at regular intervals (weekly or two-weekly), so that both they, and up to three additional family members, will be able to eat at least 4 servings per week of chicken meat, and at least 4 eggs weekly over the 4 month study period. The chicken-meat will be delivered frozen, and the eggs will be delivered refrigerated.

MEASUREMENT OF RED CELL AND PLASMA LEVELS OF FATTY ACIDS

Measurement of plasma and red cell levels of EPA, DPA and DHA will be performed at a laboratory with specific expertise in lipid analyses. Total lipids will be extracted from plasma and red cells using a modified Folch method. Phospholipids will be separated from neutral lipids by 1-dimensional thin-layer chromatography. Fatty acid methyl esters will be prepared by direct transesterification and separated using gas chromatography-mass spectrometry allowing quantification of 28 distinct fatty acid peaks. Plasma levels of omega-3-PUFAs will be expressed in microgram/gram, and red cell levels as a percentage of total fatty acids in erythrocyte membranes. The erythrocyte or red cell omega-3 index is calculated as the sum of EPA and DHA expressed as percentage of total fatty acids in erythrocyte membranes.

STATISTICAL ANALYSIS

Analyses and Reporting The study will be analyzed on an intension to treat basis. Standard summary statistics (mean, standard deviation, median, range, %) will be used to describe baseline characteristics of the participants.

Repeated measures ANOVA will be used to compare the 2 study groups. The study will be reported in accordance with the CONSORT (Consolidated Standards of Reporting Trials) 2010 statement.

Sample Size Considerations The primary end point will be the change in red cell omega-3-index at 4 months. In previous studies, the standard deviation of repeated measures of the erythrocyte omega-3 index has been found to be 0.5%. Hence with 80 participants, the study will have in excess of 95% power to detect a difference of 1% in the change from baseline in the omega-3 index between those eating enriched foods versus those eating control foods, at a 2-sided alpha-level of 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥ 18 years and < 70 years)
* Regular consumers (≥ 4 portions weekly) or willing to be regular consumers of chicken-meat.
* Regular consumers (≥ 4 eggs weekly) or willing to be regular consumers of eggs.
* Able to give informed consent.

Exclusion Criteria:

* Concurrent or recent (within last 3 months) regular intake of long-chain omega-3-PUFA supplements (containing EPA, DPA and/or DHA).
* Previous diagnosis of;

  * significant cardiovascular disease (e.g. myocardial infarction, coronary intervention, or stroke),
  * significant mental ill-health (e.g. major depression, psychosis or dementia) or
  * a haemoglobinopathy such as sickle cell anaemia or thalassemia .
* Any other serious medical condition that may adversely affect the patient's safety, limit the subject's ability to participate in the study, comply with follow-up requirements or impact the scientific integrity of the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the red cell omega-3 index at 4 months | 4 months (16 weeks)
  The difference between the red cell omega-3 index at baseline and at 4 months. The red blood cell omega-3 index is calculated as the sum of EPA and DHA expressed as a percentage of total fatty acids in erythrocyte (red cell) membranes.

SECONDARY OUTCOMES:
Change in red cell EPA | 4 months (16 weeks)
  The difference between red cell levels of eicosapentaenoic acid (EPA) at baseline and at 4 months
Change in red cell DPA | 4 months (16 weeks)
  The difference between red cell levels of docosapentaenoic acid (DPA) at baseline and at 4 months
Change in red cell DHA | 4 months (16 weeks)
  The difference between red cell levels of docosahexaenoic acid (DHA) at baseline and at 4 months
Change in plasma EPA | 4 months (16 weeks)
  The difference between plasma levels of eicosapentaenoic acid (EPA) at baseline and at 4 months
Change in plasma DPA | 4 months (16 weeks)
  The difference between plasma levels of docosapentaenoic acid (DPA) at baseline and at 4 months
Change in plasma DHA | 4 months (16 weeks)
  The difference between plasma levels of docosahexaenoic acid (DHA) at baseline and at 4 months

OTHER OUTCOMES:
A comparison of baseline plasma and red cell levels of EPA, DPA and DHA, amongst Saudi residents who regularly consume oily fish with those that do not regularly consume oily fish. | Baseline
  A comparison of baseline plasma and red cell levels of EPA, DPA and DHA, amongst Saudi residents who regularly consume oily fish with those that do not regularly consume oily fish.
An assessment of whether the plasma and red cell omega-3 index responses to the omega-3-PUFA enriched foods differs between those that do, and those who do not, include oily fish in their weekly diet. | 4 months (16 weeks)
  An assessment of whether the plasma and red cell omega-3 index responses to the omega-3-PUFA enriched foods differs between those that do, and those who do not, include oily fish in their weekly diet.

CONTACTS AND LOCATIONS:
Overall Officials: Salwa Albar, BSc, PhD, Principal Investigator — King Abdulaziz University; Alice V Stanton, MB, PhD, Principal Investigator — Royal College of Surgeons in Ireland
Locations (1):
- Department of Food Science and Nutrition, King Abdulaziz University, Jeddah, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
All de-identified individual participant data that underlie the results in a published paper, and applicable supporting clinical trial documents, may be available upon request,
Supporting Information: Study Protocol, ICF, CSR
Time Frame: 6 months after the publication of the results for each outcome.
Access Criteria: Formal requests from qualified scientific and medical researchers will be considered. Access must be consistent with the principle of safeguarding study participant privacy and consistent with the provision of informed consent.